CLINICAL TRIAL: NCT03389321
Title: A Single-center, Open-label, One-sequence, Two-treatment Study to Investigate the Effect of Macitentan at Steady State on the Pharmacokinetics of Riociguat in Healthy Male Subjects
Brief Title: Clinical Study to Investigate Effect of Macitentan on Riociguat Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AC-055-123; 2017-003502-41 (EudraCT Number)
Record Dates: First submitted 2017-12-27; First posted 2018-01-03 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Healthy Subjects
Keywords: pharmacokinetics; macitentan; riociguat
MeSH Terms: interventions — riociguat; macitentan

STUDY DESIGN:
Intervention Model Description: All the subjects included in the study will be included in a single group and will receive the drugs according to the same sequence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment A-B (Experimental): All subjects will receive treatment A followed by treatment B. Treatment A consists of a single oral dose (1 mg) of riociguat (Adempas) on Day 1. Treatment B consists of a loading oral dose of 30 mg macitentan (Opsumit) (3 tablets of 10 mg) on Day 5, then 10 mg of macitentan once daily from Day 6 to Day 15, with a concomitant administration of riociguat (1 mg) on Day 10.
  Interventions: Drug: Riociguat (Adempas); Drug: Macitentan (Opsumit)

INTERVENTIONS:
Drug: Riociguat (Adempas) — Riociguat film-coated tablets for oral administration at a strength of 1 mg
Drug: Macitentan (Opsumit) — Macitentan film-coated tablets for oral administration at a strength of 10 mg
  Other Names: ACT-064992

SUMMARY:
Both macitentan and riociguat are indicated in the treatment of pulmonary arterial hypertension (PAH) and may be administered concomitantly. The primary objective of this study is to evaluate the effect of macitentan administered for 11 days on the pharmacokinetics (PK) (i.e., amount and time of presence in the blood of riociguat) of a single dose of riociguat in healthy male subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Male subjects aged between 18 and 45 years (inclusive) at screening who signed informed consent prior to any study-mandated procedure;
* Healthy on the basis of physical examination, cardiac evaluations (12-lead ECG) and laboratory tests performed at screening;
* Body mass index of 18 to 30 Kg/m2 (inclusive) at screening;
* Systolic blood pressure 100-145 mmHg, diastolic blood pressure 50-90 mmHg, and pulse rate 50-90 beats per minute (inclusive).

Key Exclusion Criteria:

* Known allergic reactions or hypersensitivity to macitentan, riociguat, any drug of the same classes, or any of their excipients;
* Any contraindication for riociguat treatment;
* Known hypersensitivity or allergy to natural rubber latex;
* Previous history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions;
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism, or excretion of the study treatments;
* Previous treatment with any prescribed medications (including vaccines) or over the counter (OTC) medications (including herbal medicines such as St John's Wort, homeopathic preparations, vitamins, and minerals) within 3 weeks prior to first study treatment administration;
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Other protocol defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) from zero to infinity [AUC(0-inf)] of riociguat | Day 1 (pre-dose to 96 hours post-dose ), Day 10 (pre-dose to 144 hours post-dose)
  AUC(0-inf) of riociguat will be assessed following administration of riociguat alone or concomitantly with macitentan.
Maximum plasma concentration (Cmax) of riociguat | Day 1 (pre-dose to 96 hours post-dose ), Day 10 (pre-dose to 144 hours post-dose)
  The maximum observed plasma concentration of riociguat will be assessed following administration of riociguat alone or concomitantly with macitentan.

SECONDARY OUTCOMES:
Time to reach Cmax (tmax) of riociguat and its metabolite M1 | Day 1 (pre-dose to 96 hours post-dose ), Day 10 (pre-dose to 144 hours post-dose)
  The maximum observed time to reach Cmax of riociguat and M1 will be assessed following administration of riociguat alone or concomitantly with macitentan.
Elimination half life (t1/2) of riociguat and its metabolite M1 | Day 1 (pre-dose to 96 hours post-dose ), Day 10 (pre-dose to 144 hours post-dose)
  t1/2 of riociguat and M1 will be assessed following administration of riociguat alone or concomitantly with macitentan.
AUC(0-t) of riociguat and its metabolite M1 | Day 1 (pre-dose to 96 hours post-dose ), Day 10 (pre-dose to 144 hours post-dose)
  AUC(0-t) is the area under the plasma concentration-time curve from zero to time t of the last measured concentration above the limit of quantification. It will be determined for both riociguat and its metabolite M1 following administration of riociguat alone or concomitantly with macitentan.
AUC(0-inf) of riociguat metabolite M1 | Day 1 (pre-dose to 96 hours post-dose ), Day 10 (pre-dose to 144 hours post-dose)
  AUC(0-inf) of M1 will be assessed following administration of riociguat alone or concomitantly with macitentan.
Maximum plasma concentration (Cmax) of riociguat metabolite M1 | Day 1 (pre-dose to 96 hours post-dose ), Day 10 (pre-dose to 144 hours post-dose)
  The maximum observed plasma concentration of M1 will be assessed following administration of riociguat alone or concomitantly with macitentan.
Trough concentration (Ctrough) of macitentan and its metabolite ACT-132577 | Day 10 to Day 15 (before macitentan administration) and in the morning of Day 16
  Ctrough of macitentan and its metabolite ACT-132577 will be assessed during the treatment period with macitentan (Day 10 to Day 15)

CONTACTS AND LOCATIONS:
Overall Officials: Shirin Bruderer, PhD, Study Director — Actelion
Locations (1):
- CRS Clinical Research Services Mannheim, Mannheim, Germany